CLINICAL TRIAL: NCT04997122
Title: Assessment of the Health Effects of Olive Pomace Oil in Healthy and at Risk Consumers
Brief Title: Health Effects of Consuming Olive Pomace Oil
Acronym: ORUJOSALUD-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Ciencia y Tecnología de Alimentos y Nutrición (Other Government)
Responsible Party: Principal Investigator, Raquel Mateos, Principal Investigator, Instituto de Ciencia y Tecnología de Alimentos y Nutrición
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 20175429
Record Dates: First submitted 2021-08-04; First posted 2021-08-09 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Healthy; Hypercholesterolemia
Keywords: Olive pomace oil; Lipaemia; Glucose homeostasis; Inflammation; Oxidative stress biomarkers; Endothelial function
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Inflammation

STUDY DESIGN:
Intervention Model Description: After a 3-week run-in, healthy and at risk (hypercholesterolemic) volunteers were randomly allocated to one of each arm.
  Eas intervention stage lasted 4 weeks and was separated fy a 3-week wash-out.
Who Masked: Participant
Masking Description: Oils were provided in unlabelled bottles (only differed in the colors of stoppers)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olive pomace oil (Experimental): Intake of 45 g/d of olive pomace oil as the only source of oil in the diet
  Interventions: Other: Olive pomace oil
- High-oleic sunflower oil (Active Comparator): Intake of 45 g/d of high-oleic sunflower oil as the only source of oil in the diet
  Interventions: Other: High oleic acid sunflower oil

INTERVENTIONS:
Other: Olive pomace oil — Volunteers consumed during 4 weeks 45 g/d of olive pomace oil as the only source of dietary fat, used for cooking, salad dressing, toasts, etc.
  Other Names: OPO
  Arms: Olive pomace oil
Other: High oleic acid sunflower oil — Volunteers consumed during 4 weeks 45 g/d of oleic acid-rich sunflower oil as the only source of dietary fat, used for cooking, salad dressing, toasts, etc.
  Other Names: HOSO
  Arms: High-oleic sunflower oil

SUMMARY:
Healthy and at risk (hypercholesterolemic) subjects consumed during 4 weeks 45 g/d of either olive pomace oil (OPO) or high oleic acid sunflower oil (HOSO) as the only dietary fat in a randomized, crossover trial. The effects on blood lipids, glucose homeostasis, endothelial function, inflammatory cytokines, oxidative stress biomarkers and anthropometry were measured.

DETAILED DESCRIPTION:
This is the first study on the potential health effects of consumption of olive pomace oil.

After a 3-weeks run-in, 34 healthy and 30 hypercholesterolemic subjects were randomized to consume either OPO or HOSO (45 g/d) during 4 weeks, followed by a 3-week wash-out during which volunteers consumed the same amount of normal sunflower oil. During all the study, other dietary sources of fat (oil, nuts, butter, etc.) were restricted. Food intake was monitored by 3-d food records in each intervention stage and volunteers were instructed to maintain their normal physical and dietary habits (except for the changes in the consumption of other oils and fats).

At the beginning and end of each intervention stage, blood and urine samples were obtained, and blood pressure and anthropometric measurements were performed. A complete batch of analysis were performed, including serum lipids, endothelial function (flow mediated dilation (FMD), endothelial nitric oxide synthase (eNOS), vascular (VCAM-1) and intercellular (ICAM-1) cell adhesion molecules, E- and P-selectins), inflammatory and anti-inflammatory cytokines, glucose homeostasis/insulin resistance, antioxidant status and biomarkers of lipid oxidation (malondialdehyde (MDA), LDLox, ferric reducing antioxidant power (FRAP), oxygen radical absorbance capacity (ORAC), ABTS (2,2'-azino-bis(3-ethylbenzothiazoline-6-sulfonic acid) quenching capacity) and anthropometry, along with determination of incretins, adipokines, and other clinical and hematological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (Total cholesterol < 200 mg/dL; LDL-cholesterol < 135 mg/dL)
* Hypercholesterolemic volunteers (Total cholesterol 200-300 mg/dL; LDL-cholesterol 135-175 mg/dL)

Exclusion Criteria:

* BMI > 30 Kg/m2
* Smokers
* Vegetarians
* Pregnant women
* Medication/consumption of vitamins, dietary supplements
* On antibiotic treatment 3 months before starting the study
* Digestive disorders/pathologies (gastric ulcer, Chron's disease, inflammatory bowel syndrome, etc.)
* Food allergies/intolerances

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
Blood lipids | 4 weeks
  Changes on total or LDL-cholesterol levels or triglycerides in at risk (hypercholesterolemic) subjects. No effect on blood lipids expected in healthy (normocholesterolemic ) volunteers

SECONDARY OUTCOMES:
Endothelial function | 4 weeks
  Changes in the levels of selectins, adhesion molecules or eNOS levels in volunteers
Blood pressure | 4 weeks
  Changes in systolic/diastolic blood pressure in volunteers
Glucose homeostasis | 4 weeks
  Modification of fasting blood glucose or insulin levels, decrease in glycosylated hemoglobin (Hb1Ac), homeostasis model assessment (HOMA) of insulin resistance (HOMA-IR) or beta-cell function (HOMA-beta)
Inflammation | 4 weeks
  Changes in pro-inflammatory cytokines/C-reactive protein (CRP) levels
Oxidative status | 4 weeks
  Modification in serum antioxidant capacity (FRAP, ABTS, ORAC) and/or decreased levels of biomarkers of lipid oxidation (MDA, LDLox)

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Mateos, Dr, Principal Investigator — ICTAN-CSIC
Locations (1):
- Instituto de Ciencia y Tecnología de Alimentos y Nutrición, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Ramila S, Sarria B, Seguido MA, Garcia-Cordero J, Mateos R, Bravo L. Olive pomace oil can improve blood lipid profile: a randomized, blind, crossover, controlled clinical trial in healthy and at-risk volunteers. Eur J Nutr. 2023 Mar;62(2):589-603. doi: 10.1007/s00394-022-03001-y. Epub 2022 Sep 24. PMID 36153442